CLINICAL TRIAL: NCT00142597
Title: Mechanisms of Acupuncture Analgesia
Brief Title: Effectiveness of Acupuncture in Relieving Pain Due to Fibromyalgia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Richard Harris, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K01AT001111-01 (NIH); K01AT001111-01 (NIH); 1K01AT001111-01 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: acupuncture; analgesia; pain; fibromyalgia; fMRI; PET
MeSH Terms: conditions — Fibromyalgia; Agnosia; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Traditional Acupuncture (Active Comparator): Acupuncture sites will be used for active intervention.
  Interventions: Device: Acupuncture
- Sham Treatment (Sham Comparator): Sham acupuncture is used.
  Interventions: Other: Sham treatment

INTERVENTIONS:
Device: Acupuncture — Involves the insertion and manual stimulation of thin acupuncture needles into specific points in the body.
  Fibromyalgia participants will be randomized to receive 9 acupuncture treatments over the course of four weeks.
  All participants will be scanned twice using the fMRI scanner. The PET portion of the study is optional.
  Arms: Traditional Acupuncture
Other: Sham treatment — Fibromyalgia participants will be randomized to receive 9 sham treatments over the course of four weeks.
  All participants will be scanned twice using the fMRI scanner. The PET portion of the study is optional.
  Arms: Sham Treatment

SUMMARY:
This study will determine the effectiveness of acupuncture versus a placebo in altering brain activity and relieving pain due to fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is one of the most common rheumatic diseases, second only to osteoarthritis. It causes chronic muscle pain and fatigue. Acupuncture functions by targeting specific nerve pathways to different organs or parts of the body. Research has shown that acupuncture is effective in decreasing or eliminating people's sensitivity to pain in targeted regions. However, some believe that the reduction in pain is due to a placebo response rather than acupuncture itself. This study will use two brain-imaging techniques to determine the brain response to acupuncture versus a simulation of acupuncture, thereby assessing whether acupuncture is actually effective in relieving pain.

Participants in this single-blind study will be randomly assigned to receive either acupuncture or a placebo treatment. The placebo will consist of a simulation of acupuncture. Functional magnetic resonance imaging (fMRI) and positron emission tomography (PET) will be used to assess activity of brain mu-opioid receptors. These receptors are involved in the body's ability to perceive pain. All participants will be scanned twice using the fMRI scanner, once before any treatment sessions and once at the conclusion of all treatment sessions. Both fMRI sessions will involve applying pressure to the thumb to elicit a response in the brain in order to assess the corresponding fMRI blood oxygen level dependent (BOLD) signal and whether this activation changes after treatment intervention. Participants will then receive nine treatments of acupuncture or placebo outside the scanner over a 4-week period. The PET portion of this study is optional, and, if you elect to participate, your first treatment session will be performed in the PET scanner. After this first session, participants will have seven additional treatment sessions outside of the scanner over a 4-week period. The last session will be performed in the PET scanner to assess changes in mu-opioid receptor activity that may have occurred over the 4 weeks. A baseline visit to determine eligibility and a close-out visit at week 8 are also part of the participation schedule. It is very important that participants live within driving distance of Ann Arbor, MI due to the significant number of visits to our Center.

ELIGIBILITY:
Inclusion Criteria:

fMRI Inclusion Criteria:

* Has met American College of Rheumatology (1990) criteria for the diagnosis of fibromyalgia for at least 1 year
* Chronic pain more than 50% of days
* Willing to limit introduction of any new medications or treatments for fibromyalgia during the study
* Able to attend study visits up to three times weekly
* Right-handed
* Must be within driving distance of Ann Arbor, MI

PET Inclusion Criteria:

* Meets fMRI inclusion criteria
* Willing to refrain from alcohol intake for 48 hours prior to PET studies

Exclusion Criteria:

fMRI Exclusion Criteria:

* Knowledge that could prevent "blinding" of the participant to the study interventions (including previous acupuncture treatment)
* Presence of a known coagulation abnormality, thrombocytopenia, or bleeding diathesis that may preclude the safe use of acupuncture
* Autoimmune or inflammatory disease (in addition to fibromyalgia) that causes pain (e.g., rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease)
* Daily use of narcotic pain-relievers
* History of substance abuse
* Simultaneous participation in other therapeutic trials
* Pregnant or breastfeeding
* Current severe psychiatric illness (e.g., schizophrenia, major depression with suicidal ideation)
* Condition that may make exposure to fMRI medically inadvisable
* Any condition that may prevent satisfactory completion of the study protocol

PET Exclusion Criteria:

* Meets any of the fMRI exclusion criteria
* Current major depression
* Condition that may make exposure to PET medically inadvisable

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Harris, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Harris RE, Sundgren PC, Pang Y, Hsu M, Petrou M, Kim SH, McLean SA, Gracely RH, Clauw DJ. Dynamic levels of glutamate within the insula are associated with improvements in multiple pain domains in fibromyalgia. Arthritis Rheum. 2008 Mar;58(3):903-7. doi: 10.1002/art.23223. PMID 18311814

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Acupuncture: Acupuncture sites will be used for active intervention.
  Acupuncture: Involves the insertion and manual stimulation of thin acupuncture needles into specific points in the body.
  Fibromyalgia participants will be randomized to receive 9 acupuncture treatments over the course of four weeks.
  All participants will be scanned twice using the fMRI scanner. The PET portion of the study is optional.
- Sham Treatment: Sham acupuncture is used.
  Sham treatment: Fibromyalgia participants will be randomized to receive 9 sham treatments over the course of four weeks.
  All participants will be scanned twice using the fMRI scanner. The PET portion of the study is optional.
Period: Overall Study
Arm/Group | Traditional Acupuncture | Sham Treatment
Started | 23 (N=10 underwent PET imaging) | 23 (N=10 underwent PET imaging)
Completed | 20 (N=10 completed PET imaging) | 22 (N=10 completed PET imaging)
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Acupuncture | Sham Treatment | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.52 (12.85) | 44.87 (15.03) | 46.70 (13.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Mu-opioid Receptor Occupancy
Description: Here we report the change (post - pre) in mu-opioid receptor binding potential (BP) for the perigenual anterior cingulate. BP is a unitless measure and reflects the total maximum binding of receptors divided by the dissociation constant. BP = Bmax/Kd.
Time Frame: measured from baseline to week 5
Measure: Mean (Standard Deviation); unit: Unitless: binding potential is Bmax/Kd
Arm/Group | Traditional Acupuncture | Sham Treatment
Number analyzed (Participants) | 10 | 10
Unitless: binding potential is Bmax/Kd | 0.2352 (0.1911) | .0015 (.1197)

ADVERSE EVENTS:
Arm/Group | Traditional Acupuncture | Sham Treatment
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No